CLINICAL TRIAL: NCT00381927
Title: Effect of Counseling on Psychological Stress Amongst Women Felt to be at High Risk for Breast Cancer Development
Status: Completed | Type: Observational
Sponsor: Baystate Medical Center (Other)
Other Study IDs: 03-159
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Risk; Counseling; Prevention; Anxiety; BRCA1 mutation; BRCA2 mutation; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Physician Counseling

SUMMARY:
To evaluate 1) the extent of patient overestimation of breast cancer development risk in subjects referred to a physician-based high-risk breast clinic; 2) the ability of physician counseling to improve patient risk perception and reduce psychological distress; 3) to identify factors relevant in clinical practice associated with increased distress and risk perception.

DETAILED DESCRIPTION:
Patients referred to the Baystate Comprehensive Breast Center High-Risk Clinic wil, after giving consent, complete an intake evaluation of breast cancer risk, the patient's perceptions of breast cancer development risk, and the Brief Symptom Inventory-18. Physician history, physical and counseling then takes place, with sharing of risk estimates based on modified Gail model and Myriad tables regarding breast cancer risk and probability of BRCA1/2 mutation. After counseling, patients complete another assessment of risk perception and BSI-18, and again 2 months and 1 year post counseling. Recommendations for hormonal management and referral for formal genetic evaluation and testing will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at High-risk Clinic
* Ability to complete BSI-18 and risk perception questionnaire

Exclusion Criteria:

* Diagnosis of invasive breast cancer
* Diagnosis of ductal carcinoma in situ.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-08; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Wilson C Mertens, MD, Principal Investigator — Baystate Regional Cancer Program/Baystate Medical Center
Locations (1):
- Comprehensive Breast Center, Springfield, Massachusetts, United States